CLINICAL TRIAL: NCT04219943
Title: Conservative Versus Surgical Treatment of Impacted Femoral Neck Fracture in Patient 75 Years Old and Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20100103-02
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conservative Treatment for Impacted Femoral Neck Fracture (Experimental): Conservative Treatment for Impacted Femoral Neck Fracture
  Interventions: Procedure: Surgical Treatment for Impacted Femoral Neck Fracture

INTERVENTIONS:
Procedure: Surgical Treatment for Impacted Femoral Neck Fracture — Surgical Treatment for Impacted Femoral Neck Fracture

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of conservative treatment in treatment of patients over 75 years with impacted femoral neck fracture.

DETAILED DESCRIPTION:
The study is to compare clinical outcomes between conservative treatment, internal fixation, and hemiarthroplasty in patients over 75 years with impacted femoral neck fracture. All the 3 groups were evaluated by hip pain(visual analogue scale,VAS), hip function(Harris hip score,HHS), health related quality of life(European Quality of Life-5 Dimensions index scores, Eq-5d). All thses parameters were assessed at admission and 1-, 3-, 6- 12-, 24- and 36 months after intervention. Operation duration and blood loss were recorded. Mortality, union rate, complications and re-operation were also monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Patients >75 years old who were diagnosed with impacted femoral neck fracture with confirmation of mutual embedding and close combination of the fracture ends by CT or MRI scanning(including Garden 1 and 2 and varus impacted FNF) were eligible for the inclusion.

Exclusion Criteria:

Patients <75 years old, pathological fracture, nonimpacted or displaced fracture, unable to walk previously, avascular necrosis of femoral head, previous symptomatic hip pathology (such as arthritis), infection, a history of fracture in the studied hip, deformity of lower limb.

Ages: 75 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 36 months
  visual analog scale(0-10 scores) is for pain, 0 represent no pain, 10 score represent
Harris hip score | 36 months
  The score has a maximum of 100 points (no disability), covering pain (0-44 points), function (0-47 points), and range of motion and absence of deformity (0-9 points).
Eq-5d index scores | 36 months
  To rate current state of health on five dimensions (mobility, personal hygiene, usual activities, pain/discomfort, and anxiety/depression) with three possible responses for each item (no problem, some problem, unable/large problem). Integral formula: V=1-Constant-Mobility-Self-care-Usual activity-Pain/discomfort-Anxiety/depression-N3.

REFERENCES:
- [Derived] Wei P, Xu Y, Gu Y, Geng D, Yao Q, Wang L. Conservative vs Surgical Treatment of Impacted Femoral Neck Fracture in Patients 75 Years and Older. J Am Geriatr Soc. 2020 Oct;68(10):2214-2221. doi: 10.1111/jgs.16535. Epub 2020 May 15. PMID 32413174